CLINICAL TRIAL: NCT07362758
Title: Exploratory Study on mRNA Therapy Targeting CD19 for the Treatment of Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Xi Zhang, MD, Professor, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19 for Autoimmune diseases
Record Dates: First submitted 2026-01-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in vivo CAR-T drug based on LNP-mRNA, Escalation dose (Experimental)
  Interventions: Drug: in vivo CAR-T drug based on LNP-mRNA
- in vivo CAR-T drug based on LNP-mRNA, Extended dose (Experimental)
  Interventions: Drug: in vivo CAR-T drug based on LNP-mRNA

INTERVENTIONS:
Drug: in vivo CAR-T drug based on LNP-mRNA — in vivo CAR-T drug based on LNP-mRNA

SUMMARY:
Autoimmune diseases, such as immune thrombocytopenia (ITP), immune hemolytic anemia (AIHA), systemic lupus erythematosus (SLE), lupus nephritis (LN), idiopathic inflammatory myopathy (IIM), ulcerative colitis (UC), and systemic sclerosis (SSc), are a type of chronic disabling disease characterized by the immune system mistakenly attacking the body itself, leading to tissue damage and organ dysfunction.Autoimmune hematological diseases, especially difficult to treat autoimmune diseases, are a type of disease that is difficult to treat and has a significant impact on patients' lives. Although there are various treatment methods currently available, there are still many limitations to autoimmune sexually transmitted diseases that aim for long-term remission, and further research and breakthroughs are urgently needed.

The advent of COVID-19 vaccine has brought LNP mRNA technology into the public's view. After years of development, it not only shines brilliantly in COVID-19 vaccine, but also is widely used in the treatment and exploration of cancer, rare diseases and other fields. Lipid nanoparticles (LNP) are currently the most mature non viral delivery platform, capable of protecting mRNA from nuclease degradation, promoting intracellular uptake, and achieving efficient translation in vivo.

The core of LNP-mRNA technology targeting CD19 is to encapsulate the mRNA encoding specific proteins (such as anti-CD19 related proteins) in lipid nanoparticles and deliver them to the body through intravenous or intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of 14-70 years old (including threshold), gender not limited;
* 2. KPS score>60 points, life expectancy greater than 6 months;
* 3. Male and female patients of appropriate age must use reliable methods of contraception before entering the trial, during the research process until 30 days after discontinuation of medication; Reliable contraceptive methods will be determined by the primary researchers or designated personnel;
* 4. Those who can understand this experiment and have signed the informed consent form.
* 5. Before screening (at baseline), corresponding conditions should be met;
* 6. Indications for severe, recurrent, or refractory immune related diseases, including immune thrombocytopenia (ITP), autoimmune hemolytic anemia (AIHA), systemic lupus erythematosus（SLE），systemic sclerosis （SSc） etc., meet the corresponding inclusion criteria; For other types of diseases, researchers will assess whether they meet the inclusion requirements after fully evaluating the risks and benefits based on the patient's treatment needs.

Exclusion Criteria:

* 1) Study participants who are allergic or hypersensitive to any component of the investigational drug, including those who are allergic to messenger RNA (mRNA) vaccines or other RNA LNP products.
* 2) Merge any active infections that require antibiotic treatment and have not been controlled for at least one week prior to D1 administration.
* 3) Malignant tumors diagnosed within the first 2 years of screening are excluded, except for skin basal cell carcinoma, squamous cell carcinoma, or cervical cancer in situ that has been adequately treated.
* 4) Uncontrolled ischemic heart disease, including unstable angina within the previous 6 months of screening, or evidence of active ischemic heart disease on electrocardiogram.
* 5) New York Heart Association (NYHA) grade III-IV heart failure.
* 6) Study participants with combined active hepatitis B virus (HBV) infection [defined as surface antigen (HBsAg) positive and HBV DNA positive (detected by PCR)].
* 7) Study participants with combined active hepatitis C virus (HCV) infection (defined as HCV RNA positive (detected by PCR), regardless of anti HCV antibody status).
* 8) Human immunodeficiency virus (HIV) infection or history of HIV infection.
* 9) Study participants who tested positive for Treponema pallidum specific antibodies.
* 10) There may be active infection of Mycobacterium tuberculosis.
* 11) Women who are currently pregnant, breastfeeding, or planning to become pregnant.
* 12) Combining severe or recently (<2 months) diagnosed medical conditions, as determined by the researchers, may affect the study participants' tolerance to the study drug or their ability to complete the study process.
* 13) Received attenuated live vaccine or protein subunit vaccine within 30 days prior to the first study medication.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicity (DLT) | Within 28 days after the initial treatment
Maximum tolerated dose (MTD) or optimal biological dose (OBD) | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Efficacy evaluation: degree of disease remission | Within 24 weeks after the initial treatment
Pharmacodynamic characteristics: B cell clearance rate | Within at least 28 days after the initial treatment